CLINICAL TRIAL: NCT05177887
Title: Multicentric, Prospective Clinical Study of Traumacel PULVIS Haemostatic Powder Application With or Without the Use of Traumacel ENDO Applicator in the Post-market Surveillance Phase
Brief Title: Traumacel PULVIS and Traumacel ENDO Applicator in the Post-market Surveillance Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioster, a.s. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PMCF-29-11-20
Record Dates: First submitted 2021-12-01; First posted 2022-01-05 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Bleeding; Surgical Wound
Keywords: Oxidized cellulose; Haemostatic agent
MeSH Terms: conditions — Hemorrhage; Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Traumacel PULVIS (Experimental): Traumacel PULVIS will be poured into the bleeding area directly or using an applicator Traumacel ENDO Applicator.
  Interventions: Device: Traumacel PULVIS, Traumacel ENDO Applicator

INTERVENTIONS:
Device: Traumacel PULVIS, Traumacel ENDO Applicator — Haemostatic plant polysaccharide powder made of the oxidized cellulose with flexible applicator (38 cm).
  Other Names: Traumastem POWDER, Traumastem ENDO Applicator; EMOXICEL EMIPOL; Traumastem P

SUMMARY:
Traumacel PULVIS is a sterile absorbable haemostatic plant polysaccharide powder made of the oxidized cellulose. Traumacel PULVIS is designed to stop capillary bleeding as well as to prevent bleeding in the early post-operative stage, for example to stop capillary bleeding from resection areas of parenchymatous organs, muscles, to stop bleeding after endoscopy, mainly rectoscopic, procedures. The broadness of application allows for use in procedures performed in the standard way as well as endoscopically.

Traumacel ENDO Applicator is a single use, flexible, manual apparatus designed to deliver the absorbable haemostatic powder Traumacel PULVIS.

The main objective of this clinical study is to confirm the safety and efficacy of the medical device Traumacel PULVIS and Traumacel ENDO Applicator when used in accordance with their intended purpose.

The partial objectives are: to identify potential incompatibilities of Traumacel ENDO Applicator with other surgical instruments, in particular with different types of trocar cannulas; for both devices (Traumacel ENDO Applicator and Traumacel PULVIS) the identification and analysis of potential emerging risks; confirmation of the acceptability of the benefit-risk ratio; identification of any systematic misuse of the device or off-label use of the device in order to verify the correctness of its intended purpose.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18.
* Surgical intervention.
* Negative pregnancy test of women in fertile age.
* Diffuse soft tissue, vascular or parenchymal haemorrhage after conventional surgical haemostatic methods have not worked or are impractical (e.g. ligation, suture, compression, cauterisation).
* Informed consent.

Exclusion Criteria:

* Hypersensitivity or a known reaction to oxidized cellulose.
* Age under 18
* A severe clinical condition of the patient (e.g. associated illness, mental disorder) which, according to the investigator, could adversely affect patient safety and/or compliance with the procedures used in the study.
* The patient has participated in another clinical study involving a haemostatic product within 30 days prior to enrolment, or another such clinical study is planned during the subject's participation in the study.
* Pregnancy or lactation.
* If during the procedure itself, there was no need to use the test agent
* Application of any other topical haemostatic product prior to application of the test agent to the same site.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Time required to achieve haemostasis | 10 minutes
Number of subjects in whom haemostasis was achieved within 3 minutes after administration | 3 minutes
Number of subjects who required a surgical revision within 12 hours after the procedure for recurrent bleeding | 12 hours

SECONDARY OUTCOMES:
Degree of bleeding from target bleeding site | 10 minutes
Occurrence of adverse events | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Hradec Králové, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: No